CLINICAL TRIAL: NCT01333592
Title: A Multicenter, Open Label, Long-term Study of KAD-1229 in Type 2 Diabetes Patients Who Show Inadequate Glycemic Control With Diet, and Biguanide or DPP-4 Inhibitor Monotherapy
Brief Title: Long-term Study of KAD-1229 in Type 2 Diabetes Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kissei Pharmaceutical Co., Ltd. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KAD4301
Record Dates: First submitted 2011-04-06; First posted 2011-04-12 (Estimated); Results first posted 2014-11-24 (Estimated); Last update posted 2014-12-15 (Estimated); Status verified 2014-11

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; HbA1c; Long-term study
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — mitiglinide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- KAD-1229 (Experimental)
  Interventions: Drug: KAD-1229

INTERVENTIONS:
Drug: KAD-1229

SUMMARY:
The purpose of this study is to evaluate the long-term safety and efficacy of KAD-1229 as combination therapy with biguanide or DPP-4 inhibitor in type 2 diabetes patients who show inadequate glycemic control with diet, and biguanide or DPP-4 inhibitor monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes patients who show inadequate glycemic control with diet, and biguanide or DPP-4 inhibitor monotherapy
* Age in the 20 years or over inclusive
* HbA1c in the range of ≥ 6.5 to < 9%

Exclusion Criteria:

* Type 1 diabetes mellitus
* Patients with serious diabetic complications and other serious complications

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Primary Completion 2012-08 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Japan, Kanto Region, Chugoku Region, Kyushu Region, Japan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | KAD-1229 / DPP-4 Inhibitors | KAD-1229 / Biguanides
Started | 67 | 69
Completed | 58 | 52
Not Completed | 9 | 17

BASELINE CHARACTERISTICS:
Population: One patient in the KAD-1229 / biguanides group was excluded because of early discontinuation and no evaluable HbA1c.
Groups:
- Total: Total of all reporting groups
Arm/Group | KAD-1229 / DPP-4 Inhibitors | KAD-1229 / Biguanides | Total
Number analyzed (Participants) | 67 | 68 | 135
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (10.6) | 56.9 (11.5) | 58.6 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 18 | 39
  Male | 46 | 50 | 96
HbA1c [Mean (Standard Deviation); unit: %] | 7.47 (0.54) | 7.50 (0.66) | 7.49 (0.60)

OUTCOME MEASURES:

1. Secondary Outcome: Change From Baseline in HbA1c at 52 Weeks
Time Frame: at week 0 and week 52
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | KAD-1229 / DPP-4 Inhibitors | KAD-1229 / Biguanides
Number analyzed (Participants) | 58 | 53
percentage of HbA1c | -0.45 (0.69) | -0.28 (0.63)

2. Primary Outcome: Incidences of Adverse Events
Time Frame: 52 weeks
Measure: Number; unit: Participants
Arm/Group | KAD-1229 / DPP-4 Inhibitors | KAD-1229 / Biguanides
Number analyzed (Participants) | 67 | 69
Participants | 48 | 57

ADVERSE EVENTS:
Arm/Group | KAD-1229 / DPP-4 Inhibitors | KAD-1229 / Biguanides
Serious Adverse Events (participants affected / at risk) | 1/67 | 5/69
Other Adverse Events (participants affected / at risk) | 34/67 | 47/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | KAD-1229 / DPP-4 Inhibitors (N=67) | KAD-1229 / Biguanides (N=69)
large intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
acute myocardial infarction (Cardiac disorders) | 0 | 1
traumatic lung injury (Respiratory, thoracic and mediastinal disorders) | 0 | 1
colonic polyp (Gastrointestinal disorders) | 0 | 1
brain contusion (Injury, poisoning and procedural complications) | 0 | 1
lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
rib fracture (Injury, poisoning and procedural complications) | 0 | 1
skull fracture (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | KAD-1229 / DPP-4 Inhibitors (N=67) | KAD-1229 / Biguanides (N=69)
Bronchitis (Infections and infestations) | 2 | 8
Nasopharyngitis (Infections and infestations) | 17 | 30
Pharyngitis (Infections and infestations) | 6 | 2
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Dental caries (Gastrointestinal disorders) | 0 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Alanine aminotransferase increase (Investigations) | 0 | 5
γ-glutamyltransferase increase (Investigations) | 4 | 7
Blood urine present (Investigations) | 0 | 4
White blood cell count increase (Investigations) | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No